CLINICAL TRIAL: NCT04050371
Title: I-BrEATHe - Interactions Between Antiretrovirals And Transgender Hormones
Brief Title: Study of Truvada for HIV Pre Exposure Prophylaxis Using Daily Directly Observed Therapy to Look at Potential Interactions Between Truvada and Hormone Therapy
Acronym: I-BrEATHe
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco AIDS Foundation (Other); California HIV/AIDS Research Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A131155
Record Dates: First submitted 2019-08-05; First posted 2019-08-08 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: HIV Prevention; Transgender Health
Keywords: Pre Exposure Prophylaxis; HIV prevention; Emtricitabine, Tenofovir Disoproxil Fumarate; transgender health; transgender persons; drug combination; androgens; estrogens; drug combinations; transmen; non binary; Truvada; daily observed therapy
MeSH Terms: interventions — Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: All participants will receive Truvada for study duration and will take pills using daily observed therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TRUVADA DOT (Experimental): one tablet containing 200 mg of emtricitabine and 300 mg of tenofovir disoproxil fumarate as single dose with daily observed therapy performed either via video calling, or at study visit, for a total of 28 to 30 days
  Interventions: Drug: 200 mg emtricitabine and 300 mg tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: 200 mg emtricitabine and 300 mg tenofovir disoproxil fumarate — All study participants received daily observed therapy with FTC/TDF.
  Other Names: Truvada

SUMMARY:
Truvada (Emtricitabine or FTC and tenofovir disoproxil fumarate or TDF) has been approved for HIV prevention since 2012. Drug concentrations after receipt of oral Truvada for HIV Pre Exposure Prophylaxis (or PrEP) appeared to be lower in transgender women compared to Men who Have Sex with Men (MSM) in the iPrEx study, the landmark study of PrEP for HIV prevention. Concentrations were especially low among transgender women (TGW) reporting use of feminizing hormones. Reasons for the lower drug concentrations may be behavioral or biomedical, or a combination of both. While there are no systemic drug-drug interactions between TDF and oral contraception, there are known interactions involving these classes of medications with drug transporters that could affect drug concentrations in target tissues. Drug-drug interactions with natural estrogens and anti-androgenic agents used for gender affirming hormone therapy among transgender women have not been studied, neither have interactions between emtricitabine and female hormones. Concerns about the impact of PrEP on gender affirming hormone therapy is the main barrier for uptake of PrEP among transgender women. In addition, very little is known about TDF/FTC pharmacokinetics in transgender men using testosterone hormonal therapy. Drug-drug interactions with masculinizing hormones have never been properly investigated as trans gender men have not been formally involved in PrEP clinical trials or demonstrations projects.This small study will assess pharmacokinetic drug-drug interactions between tenofovir disoproxil fumarate/emtricitabine and cross-sex hormone therapy. The I-BrEATHe study is a substudy of the Triumph study, a culturally-relevant community-led PrEP demonstration project in transgender communities. The I- BrEATHe pharmacokinetic substudy will provide Truvada daily using directly observed therapy in 24 transgender women and 24 transgender men over a one month period, and will measure drug and hormone therapy levels in blood collected from participants.

DETAILED DESCRIPTION:
BACKGROUND The TRIUMPH study, or trans Research-Informed communities United in the Mobilization for the Prevention of HIV, is a new study responding to a pressing need for culturally-relevant community-led pre-exposure prophylaxis (PrEP) programs for transgender communities, especially for trans women of color who are most affected by the HIV epidemic. The TRIUMPH study will strive to identify the most effective PrEP service provision strategies which take into account the particular facilitators and barriers that transgender communities encounter in the health care system. To date, transgender women included in HIV prevention studies have been lumped into the larger aggregate of Men who have sex with Men (MSM) without taking into account the unique sociocultural context of transgender women. The TRIUMPH study will also include transgender men and other members of various transgender communities. The TRIUMPH project's goal is to identify the best methods to deliver PrEP safely and effectively to transgender communities while achieving the highest levels of adherence possible.

PrEP is the newest and most promising biomedical HIV prevention intervention yet developed and tested. The first clinical trial of PrEP ('iPrEx' or iniciativa Profilaxis Pre-Exposición) included MSM and transgender women who were at higher risk for HIV infection, and found that daily oral Truvada PrEP reduced the risk of HIV acquisition by 44% on an intention to treat basis. However, a sub-analysis of the iPrEx data conducted by Deutsch et al , found zero effectiveness on an intention to treat basis among the small subgroup of transwomen in the study. Further analyses revealed that the subgroup of trans women in iPrEx who were using hormones were less likely to have protective drug levels than those trans women not on hormones (OR 0.14, p<0.001). It is unclear if this difference is behavioral (less drug uptake) or biomedical (drug-drug interactions) in nature, or due to some combination of these factors, given the lack of pharmacokinetic (PK) studies testing for interactions between cross-sex hormone therapy (HT) and TDF/FTC, the active ingredients of Truvada. While there are studies of systemic drug-drug interactions between oral contraceptives and TDF, no such studies have been done with FTC, and no studies have been done with gender affirming HT, which differs from hormonal contraception in several respects. Drug-drug interactions with bioidentical 17-beta estradiol used for gender affirming hormone therapy among transgender women have not been studied.

The Interactions BEtween Antiretrovirals And Transgender Hormones, or I-BrEATHe study, is a sub study of the TRIUMPH study. I-BrEATHe will address one of the secondary aims of the TRIUMPH study which is to assess the pharmacokinetic drug-drug interactions between cross-sex HT and daily oral FTC/TDF.

Given that there are no PrEP studies to date that have specifically enrolled trans identified men, or have looked at the interactions between masculinizing HT and FTC/TDF, I-BrEATHe will enroll both transgender women and men. Transgender men report sexual rapport without condoms both vaginally and anally (range 26-60%), exhibit patterns of Sexually Transmitted Infections (STI) transmission and unwanted pregnancies. Transgender men also report use of sex for gender affirmation. Small convenience samples show that HIV prevalence is between 2- 5%. To date, there are no programs or PrEP recommendations specific for transgender men.

Overview of Previous Clinical Studies of PrEP There have been a large number of trials conducted with Truvada PrEP, including several demonstration projects. While there is no evidence to suggest that TDF/FTC interacts with commonly used feminizing or masculinizing hormone regimens, and evidence from studies of Antiretroviral (ARV) interactions with hormonal contraceptives have been reassuring, no direct study of these interactions has been conducted to date.

Our team led the only trans-specific sub analysis to date of the iPrEx randomized controlled trial (RCT) data as well as the open label extension (OLE) study, which included periodic dried blood spot (DBS) drug level monitoring. In iPrEx, gender identity data was not collected using current best practices ("two-step" method), making the identification of transgender participants in this multinational, multicultural and multilingual trial difficult. As all iPrEx participants had been assigned male sex at birth, a transgender subgroup of 339/2499 participants (14% of overall sample) was constructed comprised of the 29 (1%) who identified as women, 296 (12%) who identified as "trans", and 14 (1%) who reported use of feminizing hormones. None had undergone gender affirming genital surgery. Compared with MSM, transgender women more frequently reported transactional sex, receptive anal intercourse without a condom, or more than 5 partners in the past 3 months. Excluding those with a male identity who also used feminizing hormones, trans- and woman-identified participants were less likely to have TDF levels detected on random testing in the RCT (OR=0.39, 95% CI = 0.16 to 0.96, p=0.04). While there was no effectiveness of PrEP for transgender women on an intention-to-treat basis, none of the transgender participants who seroconverted had detectible drug levels at the time of HIV diagnosis. In comparison to MSM in the OLE, transgender participants had less time with protective drug concentrations (17% vs 35%, p<0.001) and were less likely to have concentrations indicating > 3 tablets/week (OR 0.71, 95% CI 0.49 to 1.03, p=0.07). Of the two transgender women who seroconverted during the OLE, both had drug levels below 350 fmol/punch in DBS, the level associated use of 2 tablets per week at the time of seroconversion. The lower concentrations were more likely if the transgender women used feminizing hormones.

Of the 7 clinical trials of Truvada PrEP for HIV prevention conducted to date, iPrEx is the only one with confirmed enrollment of trans women. No clinical studies or demonstration projects were conducted with transgender men.

STUDY RATIONALE The fact that concentrations of FTC/TDF were especially low among transgender women reporting use of feminizing hormones in the iPrEx study, which may reflect less PrEP use or a drug-drug interaction, is of high interest given that concerns about the impact of PrEP on gender affirming hormone therapy is the main barrier for uptake of PrEP among transgender women. While transgender men as a group have also been shown to be at elevated risk for HIV infection, no information about PrEP use and drug levels is available for transgender men since they have never been formally included in PrEP research. Therefore, there are no data on the potential effects of testosterone on FTC/TDF drug concentrations. FTC/TDF drug concentrations have emerged as strong correlates of protection in PrEP trials, accounting for the majority of the variation in PrEP benefits across trials and across individual participants in trials. For example, while oral FTC/TDF PrEP had 44% efficacy on an intention to treat basis in iPrEx, the protective effect was more than 90% among those with detectable drug and negligible among those with no detectable drug in blood.

The I-BrEATHe pharmacokinetic study of PrEP metabolites concentrations in association with feminizing and masculinizing hormones using directly observed therapy (DOT) will allow to establish whether interactions exist between these drugs. I-BrEATHe also provides an opportunity to include transgender men in PrEP research. Though transgender men are likely to be at lower risk for HIV acquisition than transgender women, the lack of available data regarding use of PrEP in transgender men must be remediated. I-BrEATHe will recruit equal numbers of transgender women who are using estradiol plus spironolactone (the most common HT regimen) and transgender men who are using testosterone. The primary aim will be to measure the intracellular active metabolites of TDF/FTC, tenofovir diphosphate (TFV-DP) and emtricitabine triphosphate (FTC-TP), levels in DBS collected after 1, 2, 3, and 4 weeks of video-observed Truvada for PrEP daily dosing, and comparing drug levels in the two groups receiving HT to previously acquired DBS drug levels data in MSM.

Risk / Benefit Assessment Oral Truvada for PrEP has been FDA approved since 2012. At this time, there is plentiful evidence to support the use of daily oral FTC/TDF in HIV-1-uninfected heterosexual biological men and women, and men who have sex with men for HIV prevention. The toxicity and tolerability of daily oral FTC/TDF in HIV-uninfected individuals have been established. Side effects that may arise in the first weeks of PrEP use -- nausea, abdominal cramping, vomiting, dizziness, headache, and fatigue usually go away without treatment interruption (see Truvada Prescribing information for more details). Known potential risks can be effectively managed by experienced PrEP providers. Participants enrolled in this study will be provided Truvada for PrEP within the confines of an established PrEP clinic, and will benefit from the expertise of trained staff. Individuals who may be susceptible to the possible nephrotoxic effect of FTC/TDF as determined by the measure of creatinine clearance (see exclusion criteria) will not be enrolled in the study. Long term effect of Truvada use (such as bone density loss or kidney dysfunction) are unlikely to occur over the course of this short study in otherwise healthy participants. Participants will be seen weekly by a clinician, and any adverse event immediately addressed, in addition participants will be interacting daily with study staff via phone, providing an opportunity to address any questions or concerns. Moreover, the daily interactions with study staff will provide support for adherence. Concerns about risks of combining gender-affirming hormone therapy and PrEP will be alleviated by trained providers with expertise in the management of both antiretroviral and hormone therapy. Guidelines for these matters will be provided by the University of California San Francisco Center of Excellence for Transgender Health.

STUDY OBJECTIVES Primary Objective To assess pharmacokinetics for daily oral FTC/TDF in transgender women and transgender men, and to determine if FTC/TDF drug concentrations are lower among transgender women who are using hormone therapy and in transgender men who use testosterone compared to historical controls in non-transgender MSM.

Secondary Objectives To determine if daily oral FTC/TDF is associated with comparable rates of adverse events (AEs) in transgender women and in transgender men compared to historical controls in non-transgender MSM.

STUDY DESIGN Study Overview This is a single center pharmacokinetic study of daily oral Truvada at the following FDA approved dose of one tablet containing 200 mg of emtricitabine (FTC) and 300 mg of tenofovir disoproxil fumarate (TDF) for PrEP using daily directly observed therapy (DOT).

The study will include 48 participants will be divided into two groups: one group will include 24 participants who currently describe their gender identity as "woman" or "transgender women", or other transfeminine spectrum identity, and the second group will enroll 24 participants who identify as "man" or "transgender man", or other transmasculine spectrum identity.

Each participant will be taking a single daily dose of study drug in DOT performed either via video calling, or at study visit, for a total study duration of 28 to 30 days (4 weeks).

Laboratory evaluations for HT (including testosterone, or estradiol) drug levels will be performed at enrolment, and after 4 weeks on study drug. Study drug levels will be monitored weekly in DBS while participants are on study.

Screening data will be reviewed to determine participant eligibility. Participants who meet all inclusion criteria and none of the exclusion criteria will be entered into the study.

The treatment regimen that will be used:

Truvada at the following FDA approved dose of one tablet containing 200 mg of emtricitabine and 300 mg of tenofovir disoproxil fumarate

Total duration of participant participation will be up to 4 weeks, plus the 28 days of screening window period between screening visit and on study daily observed therapy. Total duration of the study is expected to be 9 -10 months.

Pharmacogenetic testing Pharmacogenetics (PGx) studies the variability in drug response due to hereditary factors in populations. There is increasing evidence that individual's genetic background may impact the pharmacokinetics (absorption, distribution, metabolism and elimination) of drugs. The goal of the PGx analyses is to investigate a relationship between genetic factors and PK measures in I-BrEATHe, for example if there is potential unexpected or unexplained variation in drug levels. Blood samples collected for drug levels on DBS may be used for DNA extraction and PGx assessments. Participants will be specifically asked if they wish to participate in the genetic testing in the informed consent form.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* HIV antibody seronegative (negative HIV rapid test),
* 18 years or older,
* Has a smart phone with access to two-way video call capability,
* Willingness to be contacted for a short call every day for 4 weeks,
* Adequate renal function (creatinine clearance ≥ 60 ml/min estimated by the Cockcroft Creatinine Clearance Formula),
* Provides written informed consent,

For Transgender women:

* Male assigned sex at birth, and self-reported current gender identity as "woman" or "transgender women", or other trans-feminine spectrum identity,
* Current feminizing Hormone Therapy (HT) use for at least 6 months,

For Transgender men:

* Female assigned sex at birth, and self-reported current gender identity as "man" or "transgender man", or other trans-masculine spectrum identity,
* Current masculinizing Hormone Therapy (HT) use for at least 6 months with testosterone

Exclusion Criteria

* Expects to change or discontinue current HT use during the 4 weeks study period,
* Signs of symptoms of acute viral syndrome,
* Use of FTC or TDF in the past 90 days
* Receiving ongoing therapy with any of the following:

AntiRetroviral Therapy, including nucleoside analogs, non-nucleoside reverse transcriptase inhibitors, protease inhibitors or investigational antiretroviral agents interferon (alpha, beta, or gamma) or interleukin (e.g., IL-2) therapy, aminoglycoside antibiotics, amphotericin B, cidofovir, systemic chemotherapeutic agents, other agents with significant nephrotoxic potential, other agents that may inhibit or compete for elimination via active renal tubular secretion (e.g., probenecid), and/or other investigational agents

* Renal insufficiency documented as Creatinine Clearance < 60 ml/min
* For masculine-spectrum identifying persons, positive pregnancy test at screening
* At enrollment, has any other condition or factor that, based on the opinion of the investigator or designee, would preclude provision of informed consent; make participation in the study unsafe; complicate interpretation of study outcome data; or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — transmen, transwomen and gender non conforming
Enrollment: 48 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Grant, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco AIDS foundation, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279
- [Background] Deutsch MB, Glidden DV, Sevelius J, Keatley J, McMahan V, Guanira J, Kallas EG, Chariyalertsak S, Grant RM; iPrEx investigators. HIV pre-exposure prophylaxis in transgender women: a subgroup analysis of the iPrEx trial. Lancet HIV. 2015 Dec;2(12):e512-9. doi: 10.1016/S2352-3018(15)00206-4. Epub 2015 Nov 6. PMID 26614965
- [Background] Sevelius J. "There's no pamphlet for the kind of sex I have": HIV-related risk factors and protective behaviors among transgender men who have sex with nontransgender men. J Assoc Nurses AIDS Care. 2009 Sep-Oct;20(5):398-410. doi: 10.1016/j.jana.2009.06.001. PMID 19732698
- [Background] Reisner SL, White Hughto JM, Pardee D, Sevelius J. Syndemics and gender affirmation: HIV sexual risk in female-to-male trans masculine adults reporting sexual contact with cisgender males. Int J STD AIDS. 2016 Oct;27(11):955-66. doi: 10.1177/0956462415602418. Epub 2015 Sep 18. PMID 26384946
- [Background] Deutsch MB, Green J, Keatley J, Mayer G, Hastings J, Hall AM; World Professional Association for Transgender Health EMR Working Group. Electronic medical records and the transgender patient: recommendations from the World Professional Association for Transgender Health EMR Working Group. J Am Med Inform Assoc. 2013 Jul-Aug;20(4):700-3. doi: 10.1136/amiajnl-2012-001472. Epub 2013 Apr 30. PMID 23631835
- [Background] Escudero DJ, Kerr T, Operario D, Socias ME, Sued O, Marshall BD. Inclusion of trans women in pre-exposure prophylaxis trials: a review. AIDS Care. 2015;27(5):637-41. doi: 10.1080/09540121.2014.986051. Epub 2014 Nov 28. PMID 25430940
- [Background] Sevelius JM, Patouhas E, Keatley JG, Johnson MO. Barriers and facilitators to engagement and retention in care among transgender women living with human immunodeficiency virus. Ann Behav Med. 2014 Feb;47(1):5-16. doi: 10.1007/s12160-013-9565-8. PMID 24317955
- [Background] Reisner SL, Vetters R, White JM, Cohen EL, LeClerc M, Zaslow S, Wolfrum S, Mimiaga MJ. Laboratory-confirmed HIV and sexually transmitted infection seropositivity and risk behavior among sexually active transgender patients at an adolescent and young adult urban community health center. AIDS Care. 2015;27(8):1031-6. doi: 10.1080/09540121.2015.1020750. Epub 2015 Mar 19. PMID 25790139
- [Background] Anderson PL, Glidden DV, Liu A, Buchbinder S, Lama JR, Guanira JV, McMahan V, Bushman LR, Casapia M, Montoya-Herrera O, Veloso VG, Mayer KH, Chariyalertsak S, Schechter M, Bekker LG, Kallas EG, Grant RM; iPrEx Study Team. Emtricitabine-tenofovir concentrations and pre-exposure prophylaxis efficacy in men who have sex with men. Sci Transl Med. 2012 Sep 12;4(151):151ra125. doi: 10.1126/scitranslmed.3004006. PMID 22972843
- [Background] Hendrix CW, Andrade A, Bumpus NN, Kashuba AD, Marzinke MA, Moore A, Anderson PL, Bushman LR, Fuchs EJ, Wiggins I, Radebaugh C, Prince HA, Bakshi RP, Wang R, Richardson P, Shieh E, McKinstry L, Li X, Donnell D, Elharrar V, Mayer KH, Patterson KB. Dose Frequency Ranging Pharmacokinetic Study of Tenofovir-Emtricitabine After Directly Observed Dosing in Healthy Volunteers to Establish Adherence Benchmarks (HPTN 066). AIDS Res Hum Retroviruses. 2016 Jan;32(1):32-43. doi: 10.1089/AID.2015.0182. Epub 2015 Oct 15. PMID 26414912
- [Background] Zheng JH, Rower C, McAllister K, Castillo-Mancilla J, Klein B, Meditz A, Guida LA, Kiser JJ, Bushman LR, Anderson PL. Application of an intracellular assay for determination of tenofovir-diphosphate and emtricitabine-triphosphate from erythrocytes using dried blood spots. J Pharm Biomed Anal. 2016 Apr 15;122:16-20. doi: 10.1016/j.jpba.2016.01.038. Epub 2016 Jan 21. PMID 26829517
- [Background] Guideline on When to Start Antiretroviral Therapy and on Pre-Exposure Prophylaxis for HIV. Geneva: World Health Organization; 2015 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK327115/ PMID 26598776
- [Background] Liu AY, Vittinghoff E, Sellmeyer DE, Irvin R, Mulligan K, Mayer K, Thompson M, Grant R, Pathak S, O'Hara B, Gvetadze R, Chillag K, Grohskopf L, Buchbinder SP. Bone mineral density in HIV-negative men participating in a tenofovir pre-exposure prophylaxis randomized clinical trial in San Francisco. PLoS One. 2011;6(8):e23688. doi: 10.1371/journal.pone.0023688. Epub 2011 Aug 29. PMID 21897852
- [Derived] Grant RM, Pellegrini M, Defechereux PA, Anderson PL, Yu M, Glidden DV, O'Neal J, Yager J, Bhasin S, Sevelius J, Deutsch MB. Sex Hormone Therapy and Tenofovir Diphosphate Concentration in Dried Blood Spots: Primary Results of the Interactions Between Antiretrovirals And Transgender Hormones Study. Clin Infect Dis. 2021 Oct 5;73(7):e2117-e2123. doi: 10.1093/cid/ciaa1160. PMID 32766890
- See also: description of the parent Triumph study of which the I-BrEATHe pharmacokinetic study is a sub study — http://www.californiaaidsresearch.org/files/award-abstracts/prevention-and-linkage-to-care/triumph.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Transgender Men: Transgender men on stable testosterone regimen from the iBreathe Study
- Transgender Women: Transgender women on stable estradiol treatment from the iBreathe study.
Period: Overall Study
Arm/Group | Transgender Men | Transgender Women
Started | 24 | 24
Completed | 23 | 24
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Transgender Women: Transgender women on stable estradiol treatment.
- Transgender Men: Transgender men on stable testosterone regimen.
- Total: Total of all reporting groups
Arm/Group | Transgender Women | Transgender Men | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29 [26 to 40] | 34 [29 to 40] | 30 [27 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 24 | 24
  Male | 24 | 0 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants reported more than one category of race and ethnicity.
  Participants
    White | 16 | 11 | 27
    Black/African American | 4 | 6 | 10
    Hispanic/Latinx | 6 | 9 | 15
Gender Identity [Count of Participants; unit: Participants] — Transgender is defined as reporting a current gender that differs from the reported sex at birth.
  Participants
    Transgender women | 24 | 0 | 24
    Transgender men | 0 | 24 | 24
Weight (kg) [Median (Inter-Quartile Range); unit: kg] | 74 [68 to 100] | 75 [65 to 85] | 75 [66 to 94]

OUTCOME MEASURES:

1. Primary Outcome: Tenofovir Diphosphate Concentration in Dried Blood Spots (DBS)
Description: Tenofovir diphosphate concentration in dried blood spots at week 4
Time Frame: After 4 weeks of daily observed dosing of FTC/TDF
Measure: Median (Inter-Quartile Range); unit: fmol/punch
Arm/Group | Transgender Women | Transgender Men
Number analyzed (Participants) | 24 | 23
fmol/punch | 973.5 [708 to 1138.5] | 1078 [899 to 1181]

2. Other Pre Specified Outcome: Estradiol Concentration
Description: Estradiol concentrations in blood plasma by LC-MS/MS
Time Frame: Baseline and after 4 weeks of daily FTC/TDF
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Transgender Women | Transgender Men
Number analyzed (Participants) | 24 | 23
pg/mL
  Week 0 | 141.5 [89.5 to 253] | 24.2 [11.6 to 30.3]
  Week 4 | 116 [68.8 to 310] | 23.1 [13.2 to 30.4]

3. Other Pre Specified Outcome: Total Testosterone
Description: Total testosterone concentrations in blood plasma by LC-MS/MS
Time Frame: Baseline and after 4 weeks of daily FTC/TDF
Measure: Median (Inter-Quartile Range); unit: ng/dL
Arm/Group | Transgender Women | Transgender Men
Number analyzed (Participants) | 24 | 23
ng/dL
  Week 0 | 56.5 [35.3 to 71.9] | 559 [294 to 747]
  Week 4 | 56.7 [36.6 to 85] | 595 [383 to 845]

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Transgender Women: Transgender Women (Male sex assigned at birth).
- Transgender Men: Transgender men (Female sex assigned at birth)
Arm/Group | Transgender Women | Transgender Men
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 7/24 | 11/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transgender Women (N=24) | Transgender Men (N=24)
HIV infection (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea or soft stools (Gastrointestinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 6 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
lightheaded (General disorders) | 0 (0) | 1 (1)
Fever (Infections and infestations) | 0 (0) | 2 (2)
upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Fatigue (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Myalgias (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
PrEP dosing was directly observed while hormone replacement therapy was self-reported. Observation was 4 weeks which is less than required to achieve steady state PrEP drug concentrations, which were mathematically projected for the final analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT04050371/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT04050371/ICF_001.pdf